CLINICAL TRIAL: NCT04516200
Title: Effect of Transcranial Direct Current Stimulation on Sensory Integration and Risk of Falling in Diabetic Polyneuropathy
Brief Title: Effect of Transcranial Direct Current Stimulation on Sensory Integration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Sara Salah El-Din Abdel Megeed, principal investigator, MTI University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002000
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Diabetic Polyneuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Group 1: transcranial direct current stimulation and traditional physical therapy program Group 2: the same traditional physical therapy program
Who Masked: Participant
Masking Description: single blind masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial direct current stimulation (Experimental): Transcranial direct current stimulation will be applied to study group only . Anodal transcranial stimulation will be applied on left somatosensory cortex while the cathodal one will be applied on right supra-orbital area with frequency of 2m.A for 20 minutes.Stimulation will be applied three times per week for two months.
  Interventions: Device: transcranial direct current stimulation and traditional physical therapy program; Other: designed physical therapy program
- traditional physical therapy program (Placebo Comparator): traditional physical therapy program will be applied to both the control group and study group. It will be consist of sensory re-education training and balance training.Exercises will be applied three times per week for two months
  Interventions: Other: designed physical therapy program

INTERVENTIONS:
Device: transcranial direct current stimulation and traditional physical therapy program — Transcranial stimulation will be applied only for the study group.
  Other Names: Gymna- uniphy(phy-action 787)
  Arms: Transcranial direct current stimulation
Other: designed physical therapy program — sensory training and balance training

SUMMARY:
To determine the effect of Transcranial direct current stimulation on sensory integration and risk of falling in diabetic polyneuropathy.

DETAILED DESCRIPTION:
PURPOSE:

To determine the effect of Transcranial direct current stimulation on sensory integration and risk of falling in diabetic polyneuropathy.

BACKGROUND:

Diabetic polyneuropathy is the most prevalent chronic complication affecting 30% - 50% of diabetic patients. Diabetic polyneuropathy usually affect the peripheral, autonomic, and central nervous systems with several clinical symptoms .About 80% of the cases of DN manifest as distal symmetrical sensorimotor polyneuropathy which is responsible for cases of chronic pain; impaired sleep quality; increase of the falling risk associated with weakness and increase of the risk of extremities amputation. Transcranial direct current stimulation is neurophysiologic intervention that alters cortical excitability to enhance lower extremity somato-sensation and thus improve functional outcomes.

HYPOTHESES:

There will be no effect of Transcranial direct current stimulation on sensory integration and risk of falling in diabetic polyneuropathy

ELIGIBILITY:
Inclusion Criteria:

1 - Patient will be diagnosed as having Diabetic Polyneuropathy (DPN) and all patients have type II diabetes.

2-The age of the patients ranged from 35 to 55 years.

3-Clinically all patients suffered from glove stock hyposthesia, numbness and burning sensation and mild distal moror weakness

4-Patients have sensorymotor peripheral neuropathy according to neurophysiological study to detect sensory and motor conduction velocity to confirm diagnosis.

Exclusion Criteria:

1. History of diabetic ulcer and amputation .
2. Osteoporosis.
3. Fractures of lower limbs.
4. Gross musculoskeletal problems eg:burn.
5. Significant Scar tissue or calluses on the feet.
6. Peripheral vascular diseases (PVD) or Microcirculation problems.
7. Balance disturbance rather than diabetic peripheral neuropathy as ear problems, labrynthinitis, stroke or cerebellar problems.
8. Visual disturbance.
9. Autonomic neuropathy.
10. Advanced Osteoarthritis of lower limbs.
11. Nerve root compression (Radicuolopathy) affecting lower limbs.
12. Patients with implanted devices for pain control such as deep brain

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
sway index of sensory integration test | two months
  sway index of sensory integration test will be measured by biodex balance system

SECONDARY OUTCOMES:
risk of fall index | two months
  risk of fall index will be measured by biodex balance system

DOCUMENTS (1):
  • Informed Consent Form (2018-07-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT04516200/ICF_000.pdf